CLINICAL TRIAL: NCT04597983
Title: Effect of 8-week Intake of 2S-hesperidin on Performance, Body Composition and Biochemicals Markers in Amateur Cyclists
Acronym: HESPERFORMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Francisco Javier Martínez Noguera (Other)
Responsible Party: Sponsor-Investigator, Francisco Javier Martínez Noguera, Research study coordinator, Universidad Católica San Antonio de Murcia
Organization: Universidad Católica San Antonio de Murcia (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE091802
Record Dates: First submitted 2020-09-30; First posted 2020-10-22 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Power; Metabolic Disturbance; Change, Body Weight; Changes Fatty; Muscle Loss; Oxidative Stress; Inflammatory Response; Oxygen Deficiency; Acid-Base Imbalance; Electrolyte Disturbance
Keywords: Flavonoids; Polyphenols; Power; Endurance sports; Ergogenic aids; Inflammatory markers; Antioxidant markers; Body Composition; Ventilatory Thresholds; Nutrigenomic
MeSH Terms: conditions — Body Weight Changes; Fatty Liver; Muscular Atrophy; Hypoxia; Acid-Base Imbalance | interventions — Hesperidin

STUDY DESIGN:
Intervention Model Description: A randomized parallel study was conducted, where 40 amateur cyclists were divided into 2 groups: one group took 500 mg of 2S-hesperidin (n= 20) and the other group took 500 mg of placebo (microcellulose) (n= 20). All participants completed the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The company that performed the encapsulation of both the 2S-hesperidin and the placebo performed the randomization, therefore no one on the research team or the sponsors knew which group each study subject belonged to. The results of the randomization were sent to our laboratory after the end of the study to determine which subjects composed each group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2S-hesperidin (Experimental): This group took 500 mg (capsules) per day at breakfast of 2S-hesperidin (Cardiose®) for 8 weeks
  Interventions: Dietary Supplement: 2S-hesperidin
- Placebo (Placebo Comparator): This group took 500 mg of microcellulose (capsules) per day at breakfast for 8 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 2S-hesperidin — Cardiose® is a natural orange extract that due to its unique manufacturing process, maintains most of the natural hesperidin isomeric form (2S)
  Other Names: Cardiose®
  Arms: 2S-hesperidin
Dietary Supplement: Placebo — Microcellulose was used, this molecule was selected to avoid affecting the glycemia, as it can occur with dextrose or maltodextrin.
  Other Names: Microcellulose
  Arms: Placebo

SUMMARY:
This clinical study evaluates the effect of 500 mg of 2S-hesperidin for 8 weeks on performance (power generated in different metabolic zones), body composition (fat and muscle mass) and biochemical (antioxidant, inflammatory status) and metabolic (capillary blood in finger) markers in amateur cyclists. Our hypothesis is that chronic intake of 2S-hesperidin can improve performance (maximum power generated). To justify this hypothesis, we measured the parameters mentioned above, which could establish a cause-effect relationship between 2S-hesperidin intake and possible yield improvement.

DETAILED DESCRIPTION:
Participants

All participants were informed about the procedures and provided signed informed consent. The study was conducted according to the guidelines of the Helsinki Declaration for Human Research and the protocol was approved by the Ethics Committee/Institutional Review Catholic University of Murcia (Code: CE091802).

Study design

Cyclists were instructed to take the supplement along with breakfast and to continue their usual diet and training schedule. Subjects in both groups were instructed not to consume foods high in citrus flavonoids (grapefruit, lemons or oranges) for 5 days prior to and during the study, this was verified by diet recalls records.

Procedures

Participants visited the laboratory on seven occasions. Visit 1 consisted of a medical examination and blood extraction to determine health status. On visits 2 and 5, a 24-hr diet recall and a Wingate test were performed. On visits 3 and 6, another 24-hour diet recall was conducted, followed by an incremental test until exhaustion on a cycle ergometer. On visits 4 and 7, the 24-hour diet recall was repeated, and participants performed a rectangular test on the cycle ergometer. Prior to each testing session (visits 2, 3, 4, 5, 6 and 7), a standardized breakfast composed of 95.16 g of carbohydrates (68%), 18.86 g of protein (14%) and 11.30 g of lipids (18%) was prescribed by the sport nutritionist.

Pre and post evaluation test

Pre-intervention visits: 1,2,3 and 4 Post-intervention visits: 5,6 and 7

Visit 1:

Health status blood analysis: A general analysis will be performed both in the pre and post-supplementation period. The extraction will be done by venous via. (Fasting)

Medical examination: A clinical history of family and personal history, a resting electrocardiogram (ECG) and a medical examination (auscultation, blood pressure measurement, etc.) will be taken to certify that the person is healthy and not at risk to participate in the study. (Fasting)

Visits 2 and 5:

Resting Metabolic Rate (RMR): A resting test will be performed with the ergospirometer to determine macronutrient supply at rest and caloric expenditure. (Fasting)

Body composition by absorptiometric densitometry (DXA): A body composition test will be performed by the dual energy absorptiometric densitometry technique (X-ray), with the objective of to determine parameters of fat mass, fat-free mass and fat percentage. In addition, anthropometry was also used to determine changes in body composition (fat and muscle mass). (Fasting)

Anaerobic power and mechanical power production: After a standardized breakfast, a Wingate test was performed on a cycloergometer. Wingate test (WAnT) consisted of an all-out 30-s sprint on a cycloergometer (Monark Ergomedic 894E Peak Bike, Vansbro, Sweden). Breaking resistance was held constant at 7.5% of each individual's body mass. All participants were verbally encouraged to pedal as fast as possible during the entire sprint.

Visits 3 and 6:

Incremental step with final ramp test was performed on a cycle ergometer using a metabolic cart (Metalyzer 3B. Leipzig, Germany) to determine maximal fat oxidation zone (FatMax), ventilatory thresholds 1 (VT1) and 2 (VT2) and maximal oxygen consumption (VO2max). Participants began cycling at 35W for 2 min, increasing then by 35W every 2 min until RER>1.05, initialling then the final ramp (+35W·min-1) until exhaustion. The estimated functional threshold power (FTP) was calculated using the following equation [16]:

FTP (W) = Pmax (W) x 0.865 - 56.484.

Visits 4 and 7:

Rectangular test was performed on a cycle ergometer using the power output values resulting from the maximal test (FatMax, VT1 and VT2). Participants exercised continuously from FatMax, to VT1 and to VT2 for 10 min, without rest. Cardiorespiratory variables (VO2, VO2R, carbohydrate oxidation (CHO), fat oxidation (FAT) and cycling economy) were determined for each metabolic zones.

Urine samples

Main hesperidin metabolites were analysed in participants' urine. Urine samples, corresponding to 24 h urine collection from each participant before and after the supplementation, were frozen in liquid nitrogen after collection and thawed for its analysis.

All the data of the subjects who participated in the study were stored under a computer system with a security key. In addition, a record was also made of some of the paper data that was saved under key, and to which only the researchers of this project had access.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years,
* BMI of 19-25.5 kg·m-2
* At least 3 years of cycling experience and training for 6-12 h·wk-1

Exclusion Criteria:

* Were smokers or regular alcohol drinkers,
* Had a metabolic, cardiorespiratory or digestive pathology or anomaly,
* Had an injury in the prior 6 months
* Were supplementing or medicating in the prior 2 weeks
* Had non-normal values in the blood analysis parameters.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-09-22 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Maximum power | Throughout study completion, an average of 8 weeks
  During the incremental test until exhaustion, the power generated was measured maximum power (W)
Power generated at FatMax | Throughout study completion, an average of 8 weeks
  During the incremental test until exhaustion, the power generated was measured in FatMax (W)
Power generated at ventilatory threshold 1 (VT1) | Throughout study completion, an average of 8 weeks
  During the incremental test until exhaustion, the power generated was measured in VT1 (W)
Power generated at ventilatory threshold 2 (VT2) | Throughout study completion, an average of 8 weeks
  During the incremental test until exhaustion, the power generated was measured in VT2 (W)

SECONDARY OUTCOMES:
Fat mass | Throughout study completion, an average of 8 weeks
  Fat mass (g) was measured by densitometry and anthropometry.
Sum of 8 skinfolds | Throughout study completion, an average of 8 weeks
  By means of anthropometry, the sum of 8 skinfolds (mm) was calculated.
Muscle mass | Throughout study completion, an average of 8 weeks
  Muscle mass (g) was measured by densitometry and anthropometry
Resting metabolic rate | Throughout study completion, an average of 8 weeks
  Resting metabolic rate was measured by indirect calorimetry.
Superoxide dismutase (antioxidant marker) | Superoxide dismutase was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, superoxide dismutase (U/g Hb) was measured in venous blood.
Catalase (antioxidant marker) | Catalase was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, catalase (U/g Hb) was measured in venous blood.
Reduced glutathione (antioxidant marker) | Reduced glutathione was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, reduced glutathione (GSH) (nmol/mg protein) was measured in venous blood.
Oxidized glutathione (antioxidant marker) | Oxidized glutathione was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, oxidized glutathione (GSSG) (nmol/mg protein) was measured in venous blood.
GSSG/GSH ratio (antioxidant marker) | GSSG/GSH ratio was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, GSSG/GSH ratio (%) was measured in venous blood.
Hemoxigenase 1 (antioxidant marker) | Hemoxigenase 1 was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, hemoxigenase 1 (ng/mL) was measured in venous blood.
Thiobarbituric acid reactive substances (oxidant marker) | Thiobarbituric acid reactive substances was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, thiobarbituric acid reactive substances (TBARS) (mcm/L) ( are formed as a byproduct of lipid peroxidation) was measured to determine the oxidative state in venous blood.
Interleukin 6 (inflammatory marker) | Interleukin 6 was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, interleukin 6 (pg/ml) was measured in venous blood.
Tumor necrosis factor (inflammatory marker) | Tumor necrosis factor was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, tumor necrosis (pg/ml) was measured in venous blood.
C-reactive protein (inflammatory marker) | C-reactive protein was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, C-reactive protein (mg/L) was measured in venous blood.
Monocyte chemoattractant protein-1 (inflammatory marker) | Monocyte chemoattractant protein-1 was measured in pre, after the maximum power phase of the rectangular test and after the recovery phase in pre and post intervention (8 weeks) in both groups.
  During the rectangular test, monocyte chemoattractant protein-1 (pg/ml) was measured in venous blood.
Hemoglobin (oximetry marker) | Hemoglobin was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, hemoglobin (g/dL) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Hematocrit (oximetry marker) | Hematocrit was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, hematocrit (%) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Oxygen saturation (oximetry marker) | Oxygen saturation was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, oxygen saturation (%) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Oxygen partial pressure (oximetry marker) | Oxygen partial pressure was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, oxygen partial pressure (mmHg) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Carbon dioxide partial pressure (oximetry marker) | Carbon dioxide partial pressure was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, carbon dioxide partial pressure (mmHg) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Oxyhemoglobin (oximetry marker) | Oxyhemoglobin was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, oxyhemoglobin (%) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Carboxyhemoglobin (oximetry marker) | Carboxyhemoglobin was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, carboxyhemoglobin (%) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Deoxyhemoglobin (oximetry marker) | Deoxyhemoglobin was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, deoxyhemoglobin (%) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Methemoglobin (oximetry marker) | Methemoglobin was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, methemoglobin (%) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Total blood oxygen concentration (oximetry marker) | Total blood oxygen concentration was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, total blood oxygen concentration (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Total blood carbon dioxide concentration (oximetry marker) | Total blood carbon dioxide concentration was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, total blood carbon dioxide concentration (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Oxygen partial pressure at 50% oxygen saturation (oximetry marker) | Oxygen partial pressure at 50% oxygen saturation was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, oxygen partial pressure at 50% oxygen saturation (mmHg) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Relative physiological Shunt (oximetry marker) | Relative physiological Shunt was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, relative physiological Shunt (%) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Alveolar-arterial gradient (oximetry marker) | Alveolar-arterial gradient was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, alveolar-arterial gradient (mmHg) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Bicarbonate (metabolic marker) | Bicarbonate was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, bicarbonate (mmol/L) wasa measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Glucose (metabolic marker) | Glucose was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, glucose (mg/dL) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Lactate (metabolic marker) | Lactate was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, lactate (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
pH (metabolic marker) | pH was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, pH was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Actual base excess (metabolic marker) | Actual base excess was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, actual base excess (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Standard base excess (metabolic marker) | Standard base excess was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, standard base excess (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Sodium (metabolic marker) | Sodium was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, sodium (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Potassium (metabolic marker) | Potassium was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, potassium (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Chloride (metabolic marker) | Chloride was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, chloride (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)
Calcium (metabolic marker) | Calcium was analyzed pre, at the end of the FatMax phase, VT1, VT2, maximum power, FatMax2 and after the recovery phase of the rectangular test in pre and post intervention (8 weeks) in both groups.)
  During the rectangular test, calcium (mmol/L) was measured using capillary blood obtained from a finger prick and analyzed in a blood gas analyzer (ABL90 FLEX PLUS, Radiometer Iberica, Spain)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Emilio Alcaraz Ramón, Principal Investigator — Catholic University of Murcia
Locations (1):
- Research Center for High Performance Sport. Catholic University of Murcia, La Ñora, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No